CLINICAL TRIAL: NCT05696756
Title: Electronic Memory and Management Aid (EMMA) Web-based Training Evaluation for Older Adults Experiencing Memory Difficulties
Brief Title: Electronic Memory and Management Aid
Acronym: EMMA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Washington State University (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Principal Investigator, Maureen-Schmitter-Edgecombe, Regents Professor, Washington State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AZ190055
Record Dates: First submitted 2022-12-23; First posted 2023-01-25 (Actual); Last update posted 2023-01-25 (Actual); Status verified 2023-01

CONDITIONS: Subjective Cognitive Complaints; Mild Cognitive Impairment
Keywords: activities of daily living; memory; electronic aid; quality of life; health; time management
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Brief Clinician Motivational Support (Experimental): Participants will learn to use the EMMA app through a personalized web-based training platform with brief weekly motivational support from a clinician.
  Interventions: Behavioral: Personalized Web-based training for EMMA app; Behavioral: Motivational Interviewing: Clinician Support
- Technology Support Only (Active Comparator): Participants will learn to use the EMMA app through a personalized web-based training platform with technical support and reminders as needed.
  Interventions: Behavioral: Personalized Web-based training for EMMA app

INTERVENTIONS:
Behavioral: Personalized Web-based training for EMMA app — Participants will complete six sessions of training to support uptake and habit formation of EMMA app use with a personalized web-based training platform.
Behavioral: Motivational Interviewing: Clinician Support — Participants will receive weekly brief check-ins with clinicians to motivate and support the problem-solving and habit formation aspects of the web-based training.
  Arms: Brief Clinician Motivational Support

SUMMARY:
This study will evaluate the effectiveness of a personalized, web-based training intervention that was developed to teach use of an Electronic Memory and Management Aid (EMMA) application. The app-based system is designed to support everyday memory, daily activity management and positive health behavior engagement for older adults with subjective cognitive complaints or mild cognitive impairment. The investigators will also evaluate the degree to which a clinician is needed to oversee the uptake and utilization of the EMMA app during the web-based training intervention.

DETAILED DESCRIPTION:
Participants will be randomly assigned to one of two groups, "Technical Support Only" group (T-only group) and "Technical + Clinician Support" group (T+C group). Participants will be enrolled in the study for 6 months.

Participants who pass initial phone screening criteria will participate in a 2-3 hour neurocognitive assessment over zoom to establish baseline cognition, prior to beginning the intervention. Participants will also complete questionnaires and a real-world measure assessing daily functioning. After the initial assessment is complete, participants will be given one-month to learn to use the EMMA app by completing the self-paced intervention via the adaptive, web-based training platform, which includes six lessons. EMMA device-use will be captured throughout the study by the app itself.

A component of the self-paced, web-based intervention involves setting goals related to using the EMMA app. A clinician will monitor the training data and goals the T+C group participants make and conduct brief problem-solving and goal-refining sessions during the intervention weeks. These sessions are expected to be 10-15 minutes. To keep training on track, the T-only group will receive brief phone check-ins to monitor progression through the web-based intervention. Following training, there will no longer be any differences in the treatment of both groups, which will be monitored for an additional three months. Immediately following training and at the end of the 3 month monitoring period, all participants will complete the battery of questionnaires and answer a semi-structured phone interview. In addition, at the end of the 3 month follow-up, all participants will again complete the neurocognitive assessment and real-world measure of daily functioning.

ELIGIBILITY:
Inclusion Criteria:

* Must be age 50 or older
* Self-reporting subjective cognitive complaints (screening questions)
* Must be able to read and speak English

Exclusion Criteria:

* Cannot provide own informed consent
* Have a known medical, neurological or psychiatric diagnosis that explains current cognitive complaints (e.g., stroke)
* Cannot complete remote study protocol due to severe vision or hearing difficulties

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-01-20 (Estimated); Primary Completion 2024-05-20 (Estimated); Study Completion 2024-05-20 (Estimated)

PRIMARY OUTCOMES:
Change in EMMA app use daily interactions | continuous data collection through study completion up to 6 months
  Total daily use interactions derived from the EMMA app will provide a measure of how much the app is being used.
Change in Daily Assessment of Independent Living and Executive Skills (DAILIES) | at baseline and 6 month follow-up
  To measure participants capacity to complete instrumental activities of daily living (IADLs) at home, participants complete a series of brief tasks that resemble typical IADLs (e.g., paying utility bills, running errands, filling out a rebate form) six days a week for three weeks (total score; range 0-93; higher scores indicate better performance).
Change in Cognitive Self-efficacy Questionnaire (CSEQ) | at baseline, immediately post-training and 6 month follow-up
  Self-report measure of a participants confidence in their everyday cognitive abilities (mean score; range 0-10; higher scores represent better self-reported confidence in cognitive abilities).
Change in Patient-Reported Outcome Measurement Information System 29 general (PROMIS-29) | at baseline, immediately post-training and 6 month follow-up
  Self-report measure assessing a participants mental and physical health (T-score with mean of 50 and standard deviation of 10; higher scores represent worse symptomology)

SECONDARY OUTCOMES:
Change in Coping Self-efficacy Scale (CSES) | at baseline, immediately post-training and 6 month follow-up
  Self-report measure of coping abilities (total score; range 1-130; higher scores represent greater self-perceived coping abilities)
Change in Everyday Compensation questionnaire (Ecomp) | at baseline, immediately post-training and 6 month follow-up
  Self-report of everyday compensatory strategy use (mean score; range 0-4; higher scores represent better self-reported use of everyday compensatory strategies).
Change in Patient-Reported Outcome Measurement Information (PROMIS) System Applied Cognition | at baseline, immediately post-training and 6 month follow-up
  Self-perception of cognitive abilities (T-score with mean of 50 and standard deviation of 10; higher scores represent worse symptomology).
Change in Self-Efficacy for Appropriate Medication Use Scale (SEAMS) | at baseline, immediately post-training and 6 month follow-up
  Self-perception of medication management abilities (total score, range 13-39, higher scores are associated with greater self-efficacy for adherence to medications)

CONTACTS AND LOCATIONS:
Overall Officials: Maureen Schmitter-Edgecombe, PhD, Principal Investigator — Washington State University
Locations (1):
- Washington State University - Pullman; Study Remote, Pullman, Washington, United States

IPD SHARING:
Plan to Share IPD: No
Other researchers can request use of data